CLINICAL TRIAL: NCT03164915
Title: A Multicenter, Open-Label, Phase III Study to Evaluate the Efficacy and Safety of LIV-GAMMA SN Inj. in Primary Immune Thrombocytopenia (ITP)
Brief Title: A Clinical Study to Evaluate the Efficacy and Safety of LIV-GAMMA SN Inj. in Primary Immune Thrombocytopenia (ITP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Plasma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IVIg_ITP_III_2016
Record Dates: First submitted 2017-05-22; First posted 2017-05-24 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LIV-GAMMA SN Inj. (Experimental)
  Interventions: Biological: LIV-GAMMA SN Inj.

INTERVENTIONS:
Biological: LIV-GAMMA SN Inj.

SUMMARY:
The main purpose of this study is to assess the efficacy and safety of LIV-GAMMA SN Inj. in adult subjects with ITP. The primary objective of this study is to determine the responder rate. A response is defined as a platelet count of ≥30×10^9/L and at least a 2 fold increase of the baseline, confirmed on at least 2 separate occasions at least 7 days apart without bleeding. The secondary objectives are to evaluate the further efficacy assessments including duration of response, and the safety of LIV-GAMMA SN Inj.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ITP
* Mean screening platelet count of <30×10^9/L from 3 qualifying platelet counts performed within 14 days before the start of treatment, with no individual platelet count above 35×10^9/L.
* No other factors inducing ITP
* Stable doses of ITP active treatment must not have modified the dose in the preceding 1 month and must maintain their prestudy dose during the study.

Exclusion Criteria:

* Known for hypersensitivity reactions to blood products, intravenous immunoglobulin (IVIg) or immunoglobulin G
* Immunoglobulin A (IgA) deficiency
* Therapy with live attenuated virus vaccines 3 months before the first administration of LIV-GAMMA SN Inj.
* Administration of other investigational product 1 month before the first administration of LIV-GAMMA SN Inj.
* Administration of Rituximab 3 months before the first administration of LIV-GAMMA SN Inj.
* Treatment with anti-coagulants, which may affect the function of platelet
* Positive HIV, HBV, HCV
* 3-fold increase of ALT or AST compared to normal upper limit
* eCFR < 30mL/min/1.73m^2
* History of deep vein thrombosis (DVT) or IVIg-induced thrombotic compliances
* Hemoglobin > 10g/dL

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-10-24 (Actual); Primary Completion 2018-04-03 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Responder rate (CR or R) | 28 days
  The rate of subjects with complete response defined as cases with a platelet count ≥100×10^9/L, confirmed on at least 2 separate occasions at least 7 days apart without bleeding and response, which is defined as cases with a platelet count of ≥30×10^9/L and at least a 2 fold increase of the baseline count, confirmed on at least 2 separate occasions at least 7 days apart without bleeding

SECONDARY OUTCOMES:
The percentage of subjects with complete response (CR) | 28 days
  The percentage of subjects with CR defined as cases with a platelet count ≥100×10^9/L, confirmed on at least 2 separate occasions at least 7 days apart without bleeding
The percentage of subjects with response (R) | 28 days
  The percentage of subjects with R defined as cases with a platelet count of ≥30×10^9/L and at least a 2 fold increase of the baseline count, confirmed on at least 2 separate occasions at least 7 days apart without bleeding
Time to Response | 28 days
  The time from the start of treatment to the time of achievement of CR or R
Duration of response | 28 days
  the time from the achievement of CR or R to loss of CR or R
Bleeding | 28 days
  Bleeding assessment using ITP-BAT (bleeding assessment tool for ITP)

CONTACTS AND LOCATIONS:
Overall Officials: Jong Wook Lee, MD, Study Chair — The Catholic University of Korea
Locations (6):
- South Korea (6):
  - Busan National University Hospital, Busan
  - Bundang Seoul National University Hospital, Seongnam
  - Samsung Medical Center, Seoul
  - Severance Hospital, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul
  - Yangsan Busan National University Hospital, Yangsan